CLINICAL TRIAL: NCT03971266
Title: Precision Performance Status Assessment in Early Phase Clinical Trials
Brief Title: Movement and Fitness Trackers in Determining Performance Status
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0S-18-8; NCI-2019-02543 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-18-8 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prevention (Fitbit, PRO diary) (Experimental): Patients participant in movement assessment during 2 clinical trial visits. Patients also wear a Fitbit to track movements and complete a smartphone based PRO diary over 5-10 minutes to measure physical function, fatigue, sleep disturbance, social isolation, appetite, and body weight for up to 180 days.
  Interventions: Other: Activity Monitor; Other: Media Intervention

INTERVENTIONS:
Other: Activity Monitor — Wear a Fitbit
  Other Names: Activity Tracker; Activity Tracker Device; Physical Activity Measuring Device
Other: Media Intervention — Complete smartphone based PRO diary

SUMMARY:
This trial studies the use of movement and fitness trackers in determining performance status of patients with cancer who are taking part in early phase clinical. Movement and fitness trackers record movement and a number of different metrics such as steps, heart rate, and calories burned. The use of movement and fitness trackers can provide a more objective and precise estimate of patient performance status and help identify those most at risk for adverse events and hospitalization.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if in-office movement trackers identify those patients who are at highest risk for serious adverse events (SAEs) on early and developmental therapeutics (EDT) cancer trials.

SECONDARY OBJECTIVES:

Secondary objectives are related to outpatient activity trackers. I. To determine the association between the occurrence of SAEs and early trial termination, with baseline measurement of activity classification using outpatient activity trackers in the 7 days after screening visit.

II. To determine the association between the occurrence of SAEs and early trial termination, with the change in activity level classification between the week after screening visit and the week after the start of EDT.

III. To determine the association between the occurrence of SAEs and early trial termination, with averaged activity level classification in the first 4 weeks of the EDT.

OUTLINE:

Patients participant in movement assessment during 2 clinical trial visits. Patients also wear a Fitbit to track movements and complete a smartphone based Patient Reported Outcomes (PRO) diary over 5-10 minutes to measure physical function, fatigue, sleep disturbance, social isolation, appetite, and body weight for up to 180 days.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of cancer.
* Undergoing screening for a University of Southern California (USC)/Norris therapeutic clinical trial operated by the Early and Developmental Therapeutics Program which includes both phase I and II clinical trials.
* Owns a smartphone.
* Ability to understand and the willingness to sign a written informed consent.
* Willingness to wear sensors to track physical activity, Global Positioning System (GPS) location, and provide symptom ratings each night during the screening period of their clinical trial and 180 days after starting treatments.
* Able to read English, Spanish, or traditional Chinese to complete patient reported outcomes.
* Able to ambulate without an assistive device.

Exclusion Criteria:

* Missing lower limbs.
* Symptomatic brain metastases are excluded from this clinical trial. However, those with asymptomatic brain metastasis are permitted. It is permissible to have the patient on corticosteroids to eliminate symptoms of brain metastasis.
* Known movement disorder such as Parkinson?s disease, choreoathetoid movement disorders, essential tremor if that movement disorder is of sufficient severity to require drug therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Incidence of non-hematologic serious adverse events (SAEs) | Up to 60 days
  SAEs are the grade 3 or 4 non-hematologic toxicities based on CTCAE 4.0 and documented in each therapeutic clinical trials that participants were treated on. Logistic regression will be used to test the association of average measurements of Get-up and Go, and Kinect assessments collected from screening visit day (visit 1) and the first day of Early and Developmental Therapeutics (EDT) trial (visit 2) with the occurrence of SAEs after EDT given, especially during the first 60 days on EDT trial.

SECONDARY OUTCOMES:
The number of serious adverse events | Up to 60 days
  Will use logistic regression and correlation tests to test the association of outpatient movement ability classified based on metabolic equivalents (METS) collected from the first 7 days after visit 1 (baseline measurement) with the occurrence of SAEs after EDT given, and early trial determination; the correlation of activity hours and METS in the first 7 days after Visit 1 with number of SAEs observed will be tested.
The probability of early trial discontinuation as determined by withdrawal from therapy | Up to 30 days
  Early termination is defined as cancer treatment discontinued within the first 30 days of EDT trial.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge J Nieva, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California